CLINICAL TRIAL: NCT04351997
Title: Early and Delayed Cord Clamping in Infants Born by 'Two-step' Vaginal Delivery
Brief Title: Delayed Cord Clamping in Infants Born by 'Two-step' Vaginal Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Policlinico Abano Terme (Other)
Responsible Party: Principal Investigator, Vincenzo Zanardo, Professor, Policlinico Abano Terme
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 3158/AT/14
Record Dates: First submitted 2020-03-28; First posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Placental Transfusion; Hematocrit Anemia
Keywords: Placental transfusion; Two-step delivery; Early cord clamping; Delayed cord clamping
MeSH Terms: conditions — Fetofetal Transfusion | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Intervention Model Description: The investigators conducted a randomized controlled trial (RCT) ,(parallel group study wit(h 1:1 randomisation) comparing early cord clamping( ECC) (at 60 seconds) and delayed cord clamping DCC) (at 180 seconds) in 90 cases of normal birth by' two-step' delivery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early cord clamping (Experimental): Cord clamping at 60 seconds after birth.
  Interventions: Procedure: Cord clamping
- Delayed cord clamping (Experimental): Cord clamping at 180 seconds after birth,
  Interventions: Procedure: Cord clamping

INTERVENTIONS:
Procedure: Cord clamping — Umbilical cord clamping after delivery.

SUMMARY:
The investigators conducted a RCT (parallel group study with 1:1 randomisation) comparing ECC (at 60 seconds) and DCC (at 180 seconds) in 90 cases of normal birth by' two-step' delivery. In term infants born by' two-step' delivery, DCC results is a higher blood volume in the newborn and facilitates the maternal-placental-fetal exchange of circulating compounds, without potentially detrimental neonatal outcomes.

DETAILED DESCRIPTION:
Introduction: Placental transfusion supports an important blood transfer to the neonate, promoting a more stable and smooth transition from fetal to extra-uterine life with the potential to prevent iron deficiency in young children. Several studies have demonstrated that cord clamping timing is greatly relevant for facilitate placental transfusion, the transfer of extra blood from the placenta to the infant in the third stage of labor. Therefore, during natural 'two-step' delivery umbilical cord management may play a relevant role on blood passage to the neonate and it may affect neonatal hematological values and placental transfusion. The most effective way to manage umbilical cord in in 'two-step' delivery remains to be established.

Objective: The aim of the present study is to evaluate the effect of two different methods of umbilical cord management (Early Cord Clamping - ECC vs. Delayed Cord Clamping - DCC) on the placental transfusion, defined by in two-step delivery, by ∆ haematocrit (Hct) from arterial cord blood at birth and capillary blood at 48 h of age. Accounting for physiological body weight decrease. Secondary outcomes included contemporary estimate of blood gases, lactate, and glucose concentrations in arterial cord blood gas analysis.

Material and methods: This is a randomized clinical trial on the effect of different cord management newborns born by 'two-step' delivery. After obtaining parental consent, all mothers > 38 weeks' gestation will be assigned to either ECC or DCC group in a 1:1 ratio according to a randomized sequence generated by an opened, sealed, numbered, opaque envelope containing the cord clamping interventions allocation, ECC (at 1 minute) or DCC (at 3 minutes after delivery).

ELIGIBILITY:
Inclusion Criteria:

Vaginal delivery Gestational age >37 weeks Natural process of labor

Exclusion Criteria:

Cesarean section Fetal distress Major isoimmunisation Ccongenital diseases Cord abnormalities.

Ages: 2 Days to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Placental transfusion | Second day of life
  We compared the effects of ECC and DCC on placental transfusion in two-step delivery, by ∆ haematocrit (Hct) from arterial cord blood at birth and capillary blood at 48 h of age.

SECONDARY OUTCOMES:
Arterial cord blood gas analysis. | Second day of life.
  Estimate of blood gases, lactate, and glucose concentrations in arterial cord blood gas analysis.
Neonatal body weight decrease. | First and second day of life
  Neonatal body weight (Kg) and weight at discharge (Kg)
Blood gases | At birth
  pH (units)
Lactate | At birth
  mmol/L
Glucose | At birth
  mg%

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Policlinico Abano Terme, Abano Terme, Padua
  - Policlinico Abano Terme, Abano Terme
  - Padua University Hospital, Padua

IPD SHARING:
Plan to Share IPD: No
No: There is not a plan to make IPD available.